CLINICAL TRIAL: NCT03929770
Title: The Effect of Pause at the Right Ventricle on Success Rate of Final Placement in Swan-Ganz Catheterization
Brief Title: Swan-Ganz Catheter Insertion
Acronym: SG cath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2019-14
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Swan-Ganz Catheter Insertion
Keywords: Swan-Ganz catheter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with pause (Active Comparator): When the practitioner or expert investigator recognize that the tip of Swan-Ganz catheter arrive in the right ventricle, the practitioner pause the advancement for 10 sec. Next, the practitioner re-advance it to the pulmonary artery.
  Interventions: Procedure: with pause
- without pause (Experimental): When the practitioner or expert investigator recognize that the tip of Swan-Ganz catheter arrive in the right ventricle, the practitioner advance it continuously without pause to the pulmonary artery.
  Interventions: Procedure: without pause

INTERVENTIONS:
Procedure: with pause — When the practitioner or expert investigator recognize that the tip of Swan-Ganz catheter arrive in the right ventricle, the practitioner pause the advancement for 10 sec. Next, the practitioner re-advance it to the pulmonary artery.
  Arms: with pause
Procedure: without pause — When the practitioner or expert investigator recognize that the tip of Swan-Ganz catheter arrive in the right ventricle, the practitioner advance it continuously without pause to the pulmonary artery.
  Arms: without pause

SUMMARY:
The goal of this prospective randomized controlled study is to investigate the effect of pause of advancement of the Swan-Ganz catheter, which is to check whether the Swan-Ganz catheter arrive exactly at the right ventricle or not, on success rate of final placement and required time in Swan-Ganz catheterization.

The question which the investigators are trying to answer is: Continuous advancement of Swan-Ganz catheter without intended pause in the right ventricle to check whether the Swan-Ganz catheter arrive exactly at the right ventricle will decrease the trial number and required time to success final placement of Swan-Ganz catheter?

DETAILED DESCRIPTION:
Many clinicians pause advancement of Swan-Ganz catheter to check whether the Swan-Ganz catheter arrive exactly at the right ventricle or not.

The hypothesis of this study is that the intended pause during advancement of Swan-Ganz catheter in the right ventricle induce failure in advancing of it into the pulmonary artery, and that it increase the required time for final placement of it into the pulmonary artery.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need to Swan-Ganz catheterization for heart surgeries

Exclusion Criteria:

* Who doesn't agree to enroll
* Who has thrombus in the heart or the vena cavas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-04-29 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
trial number (n) | during Swan-Ganz catheterization procedure
  trial number to success placement of Swan-Ganz catheter placement into the pulmonary artery.
Success rate (%) | during Swan-Ganz catheterization procedure
  Success rate in placement of Swan-Ganz catheter placement into the pulmonary artery
required time (seconds) | during Swan-Ganz catheterization procedure
  total time to success Swan-Ganz catheter placement into the pulmonary artery

SECONDARY OUTCOMES:
incidence of arrhythmia (n) | during Swan-Ganz catheterization procedure
  incidence of arrhythmia due to Swan-Ganz catheterization
direction of placement of Swan-Ganz catheter (n) | during Swan-Ganz catheterization procedure
  direction of placement of Swan-Ganz catheter between the right pulmoary artery and the left pulmonary artery

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Boramae Hospital, Seoul, South Korea